CLINICAL TRIAL: NCT03802019
Title: The Effects of Cigarette Package Color on Smoking Behavior, Exposure and Risk Perception When Using Low Nicotine Content Cigarettes
Brief Title: Cigarette Packaging of Low Nicotine Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Cancer Institute (NCI) (NIH); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UPCC 13019; 1U54CA229973 (NIH); 832540 (Other: University of Pennsylvania IRB number)
Record Dates: First submitted 2019-01-04; First posted 2019-01-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Smoking, Cigarette
Keywords: Smoking Behavior
MeSH Terms: conditions — Cigarette Smoking; Smoking

STUDY DESIGN:
Intervention Model Description: This project will recruit current, daily cigarette smokers to a 35-day, randomized, controlled, parallel design protocol. After a 5-day period of smoking their own preferred brand cigarettes, participants will be randomized to a 30-day experimental period when they will receive either their own preferred brand (control group), or LNC cigarettes in one of four types of packaging: standard investigational (current gray packaging); red, or blue (tobacco industry strategy); or plain packaging (tobacco control strategy), for 30 days.
Who Masked: Participant
Masking Description: Participants will be informed that they will be supplied with study cigarettes with a low nicotine content, but will be blinded to the exact nicotine content and unaware that all packages will contain the same type of low nicotine content cigarette.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Own Brand (Experimental): After completing a 5-day baseline period of smoking their own brand, participants will complete a 30-day experimental period when they will continue to receive their own preferred brand of cigarettes (i.e., control group).
  Interventions: Other: Own Brand
- LNC Cigarettes + Gray Packaging (Experimental): After completing a 5-day baseline period of smoking their own brand, participants will be randomized to a 30-day experimental period when they will receive low nicotine content cigarettes in standard investigational packaging (gray).
  Interventions: Other: LNC Cigarettes + Colored Packaging
- LNC Cigarettes + Red Packaging (Experimental): After completing a 5-day baseline period of smoking their own brand, participants will be randomized to a 30-day experimental period when they will receive low nicotine content cigarettes in red packaging.
  Interventions: Other: LNC Cigarettes + Colored Packaging
- LNC Cigarettes + Blue Packaging (Experimental): After completing a 5-day baseline period of smoking their own brand, participants will be randomized to a 30-day experimental period when they will receive low nicotine content cigarettes in blue packaging.
  Interventions: Other: LNC Cigarettes + Colored Packaging
- LNC Cigarettes + Plain Packaging (Experimental): After completing a 5-day baseline period of smoking their own brand, participants will be randomized to a 30-day experimental period when they will receive low nicotine content cigarettes in plain packaging.
  Interventions: Other: LNC Cigarettes + Colored Packaging

INTERVENTIONS:
Other: LNC Cigarettes + Colored Packaging — After completing a 5-day baseline period of smoking their own brand, participants will be randomized to a 30-day experimental period when they will receive low nicotine content cigarettes in one of four types of packaging: gray, red, blue, or plain.
  Arms: LNC Cigarettes + Blue Packaging; LNC Cigarettes + Gray Packaging; LNC Cigarettes + Plain Packaging; LNC Cigarettes + Red Packaging
Other: Own Brand — After completing a 5-day baseline period of smoking their own brand, participants will be randomized to a 30-day experimental period when they will receive their own preferred brand of cigarette (i.e., control).
  Arms: Own Brand

SUMMARY:
The purpose of this study is to examine the effect of changes in cigarette package color on smoking behaviors, harm exposure, and risk perceptions when using low nicotine content (LNC) cigarettes.

DETAILED DESCRIPTION:
This project will utilize a randomized, parallel-design trial to examine the effects of low nicotine content (LNC) cigarette packaging on smoking behaviors, harm exposure, risk perceptions, and subjective ratings of cigarettes. The investigators will aim to recruit and randomize 500 daily smokers (~250 male, ~250 female) in a 35-day protocol. After completing a 5-day baseline period of smoking their own brand, participants will be randomized to a 30-day experimental period when they will receive either their own preferred brand (control), or LNC cigarettes in one of four types of packaging: standard investigational (gray packaging); red, or blue (tobacco industry strategy); or plain packaging (tobacco control strategy). Participants will be asked to attend 5 in-person sessions at the Center for Interdisciplinary Research on Nicotine Addiction (CIRNA) on Days 0, 5, 10, 20 & 35. At Intake and Days 15, 25 and 30 participants will complete sessions with research staff remotely (i.e. by video call). Sessions will occur every 4-6 days, for a total of 5 in-person and 4 remote sessions across 35 days.

ELIGIBILITY:
Inclusion Criteria:

* Self-report smoking at least 5 non-menthol, filtered cigarettes per day for at least the last 12 months.
* Not currently undergoing smoking cessation treatment or planning to quit over the duration of the study (~5 weeks).
* Plan to live in the area for the duration of the study.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.
* Able to communicate fluently in English (i.e., speaking, writing, and reading).

Exclusion Criteria:

* Smoke menthol cigarettes greater than 20% of the time.
* Smoke cigarettes of non-standard circumference (e.g., wides, slim, capri, etc.)
* Use of any nicotine containing products other than cigarettes. Participants reporting isolated use of other nicotine containing products less than 5 times per month are eligible to participate.
* Attempt to quit smoking over the duration of the study period.
* Provide a Carbon Monoxide (CO) reading less than 5 parts per million (ppm) at Session 1 (D0).
* History of substance abuse (other than nicotine) in the past 12 months and/or currently receiving medical treatment for substance abuse. Attendance at alcoholics anonymous or narcotics anonymous meetings will not be considered medical treatment for the purposes of this protocol.
* Current alcohol consumption that exceeds 25 standard drinks/week.
* Women, including all individuals assigned as "female" at birth, who are pregnant, breast feeding, or planning a pregnancy over the duration of the study period.
* Any impairment including, but not limited to, visual, physical, and/or neurological impairments preventing the proper completion of the study procedures. Notable impairments will be evaluated on a case-by-case basis by the Principal Investigator and/or the Study Physician.
* Color blindness.
* Serious or unstable medical condition. Applicable conditions will be evaluated on a case-by-case basis by the Principal Investigator and/or the Study Physician.
* Lifetime history of schizophrenia, psychosis, and/or bipolar disorder.
* Current diagnosis of active major depression. Participants who maintain a diagnosis of major depression who have not experienced any major depressive episodes in the past 6 months and are stable on antidepressant medication(s) are eligible to participate.

Additional, general reasons for exclusion include:

* Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact subject safety, study data, and/or the study design as determined by the Principal Investigator and/or Study Physician.
* Any circumstance, medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance as determined by the Principal Investigator and/or Study Physician. Participants may be withdrawn for any of the aforementioned reasons at any point throughout the study.
* Significant non-compliance with protocol and/or study design as determined by the Principal Investigator and/or Study Physician. Participants may be withdrawn at any point throughout the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Daily Cigarette Consumption | Day 0 through Day 35
  Daily cigarette consumption will be assessed by participant self-report and verified through collection of spent filters for all cigarettes smoked throughout the entire 35-day study.
Total Puff Volume/Puff Duration | Day 0 through Day 35
  Total puff volume/puff duration (the sum of all puff volumes/duration per cigarette) will be collected for each cigarette smoked during each laboratory session using a standardized video scoring procedure. Total puff volume will be assessed for each cigarette smoked at in-person and remote sessions throughout the entire 35-day study.
Carbon Monoxide (CO) | Days 0, 5, 10, 20 and 35
  The investigators will assess CO (measured in parts per million [ppm]), a measure of toxicant exposure, at the onset of each session, as well as before and after each cigarette smoked during each in-person laboratory session. CO collected at the onset of each session represents daily exposure, while CO boost - the change in CO values before and after smoking a cigarette - estimates smoke exposure due to smoking an individual cigarette.
Total Nicotine Equivalents | Days 5 and 35
  Urine collected at Day 5 and Day 35 will be assessed for changes in total nicotine equivalents, nicotine plus its primary metabolites, across the experimental study period (Days 5-35). Total nicotine equivalents will be measured in nanograms per milliliter (ng per mL).
Total NNAL | Days 5 and 35
  Urine collected at D5 and D35 will be assessed for changes in NNAL, a biomarker of carcinogen exposure, across the experimental study period (Days 5-35). Total NNAL will be measured in nanograms per milliliter (ng per mL).

SECONDARY OUTCOMES:
Subjective Cigarette Ratings (Visual Analog Scale [VAS] of Cigarette Characteristics) | Days 0, 5, 10, 20 and 35
  Participants will provide subjective ratings of each cigarette smoked during each in-person laboratory session using a 14-item, 100 mm visual analog scale (VAS) of cigarette characteristics. Anchors are item-specific (e.g., taste: 0 = "very bad," 100 = "very good"), with lower scores indicating less favorable ratings.
Cigarette Risk Beliefs | Days 0, 5, 20, and 35
  To assess risk beliefs about the assigned cigarettes, the investigators will use an 8-item, 5-point scale (1 = definitely untrue; 5 = definitely true) including previously validated items (i.e., "Compared to your own cigarettes, the cigarettes you are currently smoking: are lower in nicotine"). The Cigarette Risk Beliefs questionnaire will be administered at Session 1 (Day 0) before the lab cigarette (18-item baseline version), Session 2 (Day 5) before lab cigarette 1 and 2, Session 5 (Day 20) before the lab cigarette, and Session 8 (Day 35) before the lab cigarette.
Cigarette Craving (Questionnaire on Smoking Urges [QSU]) | Days 0, 5, 10, 20 and 35
  Participants will report cigarette craving at the onset of each in-person session. Craving will be assessed using a summary score and two factor subscales (i.e., desire to smoke and craving due to anticipation of negative affect relief) from a 32-item Questionnaire on Smoking Urges (QSU). Participants will respond to each item along a 7-point scale (1=Strongly disagree; 7=Strongly agree).
Cigarette Withdrawal (Withdrawal Symptom Checklist [WSC]) | : Days 0, 5, 10, 20 and 35
  Participants will report cigarette withdrawal at the onset of each in-person session. Withdrawal will be assessed using a summary score from the 20-item (21 items at Session 1 [Day 0]) revised version of the Withdrawal Symptom Checklist with a one-week frame of reference (WSC-W). Specifically, participants will respond regarding to how they felt in regards to each potential withdrawal symptom along a 4-point scale (0=Not Present; 3=Severe).
Total Puff Count | Day 0 through Day 35
  Participants will be video recorded while smoking each lab cigarette in order to collect smoking topography data. During remote sessions, participants will be asked to record a video of their smoking to collect smoking topography data. We have previously used a procedure where we score digital files (video recorded) smoking sessions that has good reliability and consistency (ICCs >.55) for number of puffs taken, interpuff interval, total time lit, and amount smoked (by mass and length), and propose to quantify cigarette smoking behavior using the same procedures.
Puff Duration | Day 0 through Day 35
  Participants will be video recorded while smoking each lab cigarette in order to collect smoking topography data. During remote sessions, participants will be asked to record a video of their smoking to collect smoking topography data. We have previously used a procedure where we score digital files (video recorded) smoking sessions that has good reliability and consistency (ICCs >.55) for number of puffs taken, interpuff interval, total time lit, and amount smoked (by mass and length), and propose to quantify cigarette smoking behavior using the same procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Strasser, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research for Nicotine Addiction, Philadelphia, Pennsylvania, United States